CLINICAL TRIAL: NCT00480311
Title: WHODAS-II for Patients With Symptomatic Lumbar Spinal Stenosis
Brief Title: World Health Organization Disability Assessment Schedule II (WHODAS-II) for Patients With Symptomatic Lumbar Spinal Stenosis
Status: Terminated | Type: Observational
Why Stopped: Recruitment was so slow, that it made the study impossible. Organizational changes made it impossible for recruiting centers to continue recruitment
Sponsor: Kovacs Foundation (Other)
Responsible Party: Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation
Other Study IDs: FK-R-19
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Lumbar Spinal Stenosis
Keywords: symptomatic; lumbar spinal stenosis; disability; fear avoidance beliefs; quality of life
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Measurement characteristics of WHODAS II (World Health Organization Disability Assessment Schedule).
  Interventions: Other: WHODAS II (World Health Organization Disability Assessment Schedule II)

INTERVENTIONS:
Other: WHODAS II (World Health Organization Disability Assessment Schedule II) — To determine the measurement characteristics of WHODAS II (World Health Organization Disability Assessment Schedule).

SUMMARY:
The main purpose of this study is to determine the measurement characteristics of WHODAS-II (World Health Organization Disability Assessment Schedule II), as well as to analyze its correlation with symptomatic lumbar spinal stenosis (Visual Analog Scale, VAS), disability (Spanish version of the Roland Morris Questionnaire, RMQ), fear avoidance beliefs and attitudes (Spanish version of the FAB Questionnaire, FABQ), and quality of life (SF-12). Measurements will be taken at baseline and 6 days later (day 7).

ELIGIBILITY:
Inclusion Criteria:

* Patients seen for symptomatic lumbar spinal stenosis
* With signs of neurogenous claudication
* MRI or CAT scan concordant with observed signs
* Able to read and write
* Have signed the informed consent form

Exclusion Criteria:

* Central nervous system pathology (with or without treatment)
* Diagnosis of rheumatic inflammatory disease or fibromyalgia
* Red flags for underlying systemic disease
* Criteria for diagnosis of disc herniation
* Symptoms suggesting saddle anesthesia, cauda equina, loss of sphincter tone or paraparesis
* Motor deficit that progresses or does not improve in 6 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at Hospital Universitario Marqués de Valdecilla in Santander, Spain - for symptomatic lumbar spinal stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Measurement characteristics of WHODAS-II | At baseline and at 7 days

SECONDARY OUTCOMES:
Correlation between WHODAS-II and VAS, RMQ, FABQ and SF-12 in symptomatic lumbar spinal stenosis | At baseline and at 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, Spain; José Luis Peña, MD, Principal Investigator — Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain
Locations (1):
- Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain

REFERENCES:
- [Background] Bombardier C. Outcome assessments in the evaluation of treatment of spinal disorders. Introduction. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3097-9. doi: 10.1097/00007632-200012150-00002. No abstract available. PMID 11124723
- [Background] Chwastiak LA, Von Korff M. Disability in depression and back pain: evaluation of the World Health Organization Disability Assessment Schedule (WHO DAS II) in a primary care setting. J Clin Epidemiol. 2003 Jun;56(6):507-14. doi: 10.1016/s0895-4356(03)00051-9. PMID 12873644
- [Background] van Tubergen A, Landewe R, Heuft-Dorenbosch L, Spoorenberg A, van der Heijde D, van der Tempel H, van der Linden S. Assessment of disability with the World Health Organisation Disability Assessment Schedule II in patients with ankylosing spondylitis. Ann Rheum Dis. 2003 Feb;62(2):140-5. doi: 10.1136/ard.62.2.140. PMID 12525383